CLINICAL TRIAL: NCT04835350
Title: Feasibility Study of the Pancreas4ALL Closed-loop Automated Glycemic Control System in Patients With Type 1 Diabetes Mellitus: Pancreas4ALL Project - Good News Study - Phase I
Brief Title: Feasibility and Safety Study of the Automated Insulin Delivery Closed Loop System Pancreas4ALL
Acronym: ASAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lenka Petruzelkova (Other)
Collaborators: CLOSED LOOP Systems s.r.o. (Unknown)
Responsible Party: Sponsor-Investigator, Lenka Petruzelkova, MD, PhD, University Hospital, Motol
Organization: University Hospital, Motol (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 01-CIP-27-11-20
Record Dates: First submitted 2021-03-23; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Type 1 Diabetes
Keywords: closed loop system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Pilot prospective controlled monocentric open-label, randomized study evaluating the feasibility and safety of Pancreas4All automated "closed loop" system.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hybrid closed loop group (No Intervention): Patients using AID system Pancreas4ALL in mode hybrid closed loop.
- Closed loop meal announcment (Experimental): Patients using AID system Pancreas4ALL in mode meal announcment. They only announce what amout of carbs going to eat. They calculate no bolus
  Interventions: Device: Pancreas4ALL - meal announcement or full closed loop
- Full closed loop (Experimental): Patients using AID system Pancreas4ALL in mode full closed loop. They eating with no permission and they do not calculate and sending bolus anymore.
  Interventions: Device: Pancreas4ALL - meal announcement or full closed loop

INTERVENTIONS:
Device: Pancreas4ALL - meal announcement or full closed loop — Patient using AID Pancreas4ALL in mode meal announcment or full closed loop.
  Arms: Closed loop meal announcment; Full closed loop

SUMMARY:
Pilot prospective controlled monocentric open-label, randomized study evaluating the feasibility and safety of the Pancreas4All automated "closed loop" glycemic control system.

DETAILED DESCRIPTION:
1. Screening - day 0
2. Hospitalization (Day 1-10) Day 1 - Deployment of study equipment, patient education Day 2 - Start of study, activation of Pancreas4ALL closed loop in mode - hybrid closed loop (2.7.1) Day 4 - Randomization of patients to Group A and to Group B Group A - Activation of Pancreas4ALL closed loop in closed loop mode - "food announcement" (2.7.2) Group B - Activation of Pancreas4ALL closed loop in mode - full closed loop mode (2.7.3) Day 7 - Crossover - Group exchange Day 10 - Return to the initial treatment modality.
3. Termination of the study

Detailed description of the clinical trial - study control plan:

Outpatient check:

1. Signing of informed consents to the study and GDPR consent to the processing of personal data by the legal representative and the entity that will be included in the study
2. Urine pregnancy test for women and girls after menarche
3. Blood collection for the determination of HbA1c, TSH and creatinine
4. Evaluation of entry criteria (inclusion criteria); if all criteria are met, the subject will be included in the study.

Day 1:

1. Hospitalization in the inpatient part of the University Hospital and the 2nd Medical Faculty of Charles University, Department of Endocrinology and Diabetology.
2. Download data from an existing pump / sensor for the last 3 months to Carelink or Diasend
3. Creating a DexCom Clarity and Diasend / Tidepool account (certified patient data store)
4. Training of the patient in the use of the DANA RS Diabcare pump and the DexCom G6 CGM
5. Training of Samsung S10e mobile phone with active version of Pancreas4ALL application connected to Dana RS Diabcare and Dexcom G6 IP - mode open loop
6. Application of DANA RS Diabcare insulin pump and CGM Dexcom G6 to the patients
7. Optimization of basal dose and bolus calculator settings using Pancreas4ALL advisor (calculation based on patient's age, weight and CDD)
8. Education about the necessary inputs (data entered by the patient) into the Pancreas4ALL application.
9. Activation of the Pancreas4ALL application - open loop. Preprandial bolus calculated by the patient using a bolus calculator, part of the Pancreas4ALL application.
10. Completion of the Quality of Life (QoL) Questionnaire PedsQl

Defined Pancreas4ALL settings for all subjects.

* Target glycemia 5.5 mmol / mol
* Active insulin time 6 hours
* Setting automatic functions: In case of hypoglycemia (glycemia below 3.9 mmol / l), a temporary blood glucose target of 8 mmol / l is automatically set for 30 minutes after the hypoglycemia has occurred.

Another activities:

* In case of physical activity, it is recommended that the patient temporarily increase the target glycemia to 8 mmol / l, switch to a temporary profile of 70-80% depending on the intensity of physical activity (automatic recalculation of basal dose, insulin sensitivity, insulin carbohydrate ratio to 70-80%)
* In case of illness accompanied by an increase in glycaemia, the patient is recommended to switch to a temporary profile of 120-150% (automatic recalculation of the basal dose, insulin sensitivity, insulin carbohydrate ratio at the set 120-150%)

Day 2:

1) Initiation - activation of the "closed loop" Pancreas4All in the hybrid closed loop mode (2.7.1)

1. The patient will enter the number of carbohydrates eaten into the application, using the bolus calculator to calculate the preprandial bolus.
2. Meal blood glucose will be corrected using the Pancreas4All automated system.
3. In case of glycemia above 13 mmol / l 30 min after a meal, the correction bolus will be calculated using a bolus calculator. Hyperglycemia management see appendix.
4. In case of hypoglycaemia (glycaemia <3.9 mmol /), the subject will be given dextrose in the form of tablets or a sweet drink (the amount of dextrose will be calculated according to the patient's weight, current level and glycemic trend) See Appendix.

Day 4:

1. Randomization to group A and group B
2. Randomization will be performed using an IT application according to age, gender, weight and input glycated hemoglobin.
3. Randomization:

   1. Group A: Activation of Pancreas4ALL in closed loop mode in "meal announcement" (version 2.7.2). The patient will only enter a notification in the application that he is going to eat.
   2. Group B: Activation of the Pancreas4ALL application in mode full closed loop mode (version 2.7.3). The subject will not enter any notification or notification into the application that it is going to eat.
4. Other settings + glycemic control remain as in the previous phase.

Day 7 - Cross-over - change of settings for groups A and B:

1. The basic settings remain unchanged
2. Change the setting mode in groups A and B
3. Blood glucose control see above.

Day 10 - Visit 2 - End of study:

1. Download data from pump to DexCom clarity and Diasend / Tidepool, check data storage from IP and sensor
2. Evaluation of glycemic control for the last week
3. Completion of the PedsQl Quality of Life (QoL) Questionnaire + System Satisfaction Questionnaire.
4. Termination of the study - return to the standard treatment modality of the patients

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included in the study if they meet the following entry criteria:

1. The subject was diagnosed with type 1 DM ≥ 1 year
2. The subject is aged 15-25
3. The subject has an HbA1C value between 43 mmol / mol and 75 mmol / mol at the time of the screening visit
4. The subject must have experience with insulin pump therapy and CGM ≥ 3 months
5. The subject is willing to use the system Pancreas4ALL continuously throughout the study

Exclusion Criteria:

1. The subject does not tolerate the adhesive patch at the sensor site for CGM 2. Women of productive age who have a positive pregnance test at the time of screening or are planning to become pregnant at the time of the study 4. The subject underwent the following diagnoses in the year preceding screening: myocardial infarction, unstable angina pectoris, coronary artery bypass passage, stent insertion into the coronary artery, transient ischemic attack, cerebrovascular accident, angina pectoris, congestive heart failure, ventricular arrhythmia or thromboembolism 5. The subject has an abnormal (> 1.5x times the upper reference limit, as assessed by the laboratory) creatinine at the time of screening 6. The subject has clinically significant abnormalities (outside the reference range as assessed by the laboratory) of thyroid stimulating hormone (TSH) at the time of screening 7. The subject has taken any oral or injectable corticosteroids in the last 8 weeks prior to the screening visit, or plans to take any oral or injectable corticosteroids during the study 8. The subject is actively involved in any research study (drug or instrumental) in which he or she has undergone treatment with a research drug or research facility in the previous 2 weeks prior to the screening visit.

9. The subject is currently using illicit drugs 10. The subject is currently abusing prescription drugs 11. The subject is currently addicted to alcohol 12. The subject is taking pramlintide (Symlin) or an SGLT2 inhibitor at the time of the screening visit 13. The subject suffers from a visual impairment that does not allow him to participate in the study and to safely perform all tasks within the study, as determined by the investigator 14. The subject has planned elective surgery requiring general anesthesia for the duration of the study 15. The subject has currently been diagnosed with an eating disorder such as anorexia or bulimia 16. The subject has been diagnosed with chronic renal failure leading to chronic anemia 17. The subject is dialyzed

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
The feasibility of the prototype device Pancreas4ALL | ten days
  Percentage of time of automatic control of glucose by Pancreas4ALL would be > 90%
The safety of the prototype device Pancreas4ALL | ten days
  Percentage of time spent in hypoglycemia 2.degrees (<3 mmol / L) would be < 1% during sutomatic glucose control by Pancreas4ALL

SECONDARY OUTCOMES:
GCM parametrs of glycemic control | ten days
  Calculation of Time in range (3.9 - 10 mmol / l) which would be > 75% throughout the study Translation results "The secondary goal is excellent glycemic control in all tested versions of the Pancreas4ALL closed loop application (version 2.7.1, version 2.7.2, version 2.7.3), defined as the time spent in Time in range (3.9 - 10 mmol / l) > 70% throughout the study. "
Quality of life of patient living on closed loop system Pancreas4ALL | seven days
  PedsQL Diabetes Module 3.2 - questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lenka Petruzelkova, MD, PhD, Principal Investigator — Department of Paediatrics, Motol University Hospital, Charles University
Locations (1):
- Department of Paediatrics, Motol University Hospital 2nd Medical Faculty in Prague, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
basic characteristic of participants and all results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months

REFERENCES:
- [Derived] Petruzelkova L, Neuman V, Plachy L, Kozak M, Obermannova B, Kolouskova S, Pruhova S, Sumnik Z. First Use of Open-Source Automated Insulin Delivery AndroidAPS in Full Closed-Loop Scenario: Pancreas4ALL Randomized Pilot Study. Diabetes Technol Ther. 2023 May;25(5):315-323. doi: 10.1089/dia.2022.0562. Epub 2023 Mar 13. PMID 36826996